CLINICAL TRIAL: NCT01768234
Title: Cognitive Effects of Drinking Water and Improving Hydration Status Among Schoolchildren
Brief Title: Dehydration Among School Children- Mali
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Save the Children (Other)
Responsible Party: Principal Investigator, Matthew Freeman, MPH, PhD, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00062354
Record Dates: First submitted 2012-12-19; First posted 2013-01-15 (Estimated); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Dehydration
Keywords: cognition; hydration; schoolchildren
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supplemental water (Experimental): This arm receives up to 2 L of supplemental water during the course of the testing day.
  Interventions: Other: Supplemental water
- Control (No Intervention): No supplemental water provided

INTERVENTIONS:
Other: Supplemental water — 1-2L of supplemental water provided between pre-test and post-test
  Arms: Supplemental water

SUMMARY:
There is a large body of evidence from adult populations suggesting cognition in adults is affected by hydration status. The few studies conducted in the global North in populations of schoolchildren indicate that drinking water has an impact on pupil performance on basic cognitive tasks. No studies assessing the impact of dehydration and cognition in schoolchildren have been carried out in the global South, where access to water is the poorest and dehydration prevalence is likely higher. This study will examine the effect of drinking supplementary water during the school day on hydration status and on cognitive test scores in schoolchildren in Mali, West Africa.

The investigators hypothesize that providing supplemental water will result in a decrease in prevalence of dehydration in the study group and will result in an improved performance on cognitive test scores.

Data will be collected from up to four purposively-selected schools in the Sikasso region of Mali, from up to a total of 300 children. At each school pupils in grades 3-6 will be eligible for recruitment. Research staff will explain the study to pupils at the school and individually request informed oral assent for participation. A waiver of parental consent for pupil interviews will be secured from the Ministry of Education. At each school, school directors will be asked to sign in loco parentis ("in the place of parent") on behalf of the pupil participants.

Children that assent to participate in the study will be randomly allocated to the intervention or control group. Data collection will take place at each school over two days within a one-week period, with one study group tested on each of the two days. On the intervention testing day, all study participants will receive supplementary water. On the control testing day, no study participants will receive supplementary water. Testing procedures in both groups is identical and will include a five-minute interview, two cognitive testing sessions of 45 minutes each, and collection of two urine samples during the day. None of these activities collect personal data or identifiers, and the urine sample will not be stored.

All data collection will occur at the school and will be conducted by trained local enumerators. There are no risks to participation other than a small amount of class time missed by pupils, and great efforts will be made to minimize time outside of class.

DETAILED DESCRIPTION:
Background and Specific Aims

The purpose of this study is to evaluate the impact of improved water access on the cognitive performance and mood of primary school children in West Africa.

There is a considerable body of research assessing links between dehydration to reduction in cognitive ability and mood, but few of these studies involve children and only one such study has taken place outside of Europe. UNICEF estimates that only 47% of schools in low-income settings have access to any water during the day. Emory researchers have recently quantified the impact of improved water, sanitation, and hygiene (WASH) access in school on health and education measures. A better understanding of the impact of water intake on hydration has importance for the growing number of school-based WASH interventions in developing countries, not only for purposes of pure scientific knowledge but also for advocacy from donors and national governments.

To this purpose, the investigators have identified the following objectives:

* Refine a battery of cognitive tests for children in low-income settings;
* Assess the levels of dehydration among children in poor and arid settings;
* Quantify the effect of improved water access on hydration status and cognition; and
* Compare different field hydration assessment techniques for accuracy and ease of use

Study significance

Data collected through this research will contribute new evidence for use in school WASH intervention programming and international advocacy, as well as provide significant and groundbreaking evidence for improving water quantity in schools. There is an increasing body of evidence of the impact of improved school WASH conditions on reduced school absence, parasitic infection, and diarrheal disease. However, the precise mechanisms of improved educational attainment have yet to be fully explored. Linking drinking water availability directly to cognitive skills would provide one such explanatory mechanism.

School inclusion criteria

This study will involve children in grades 3-6 attending primary schools in Sikasso, Mali.

* No water point access within 2 km
* Within 1.5 hours drive from Bamako.
* Program activities have not commenced in the school

Setting

Data collection activities will take place at up to four primary schools. Paper cognitive tests and questionnaires will be administered by research staff to pupils inside of the classroom, under the supervision of the classroom instructor. Surveys and taking of informed assent will be conducted in a private space outside of the classroom.

Procedures for subjects

Data collection procedures will be identical on each day of data collection and will follow the general below, which may be slightly modified to account for specific school schedules.

Morning (*Denotes Day 1 activities only)

* 7:30 - 8:00 Class description of the study* (Group setting)
* 8:00 - 8:45 Pupil assent process*, screening*, interview, urine sample collection (One-by-one).

Afternoon

* 2:00 - 2:30 Urine sample collection (One-by-one)
* 2:30-3:15 Cognitive testing + self-report scales (Group setting)

Data collection activities

Pupil interview. The pupil interview will be conducted prior to collecting the morning urine sample on each group's respective testing day. It will contain questions on drinking and eating habits at school and at home. Pupils will be excused from class to complete the interview one at a time, and immediately following the interview will be asked to provide a urine sample before returning to class.

Urine sample collection. Pupils will be asked to provide one urine sample in the morning and one urine sample in the afternoon on the day of data collection for their respective group. Pupils will be provided with a urine sample container marked with a unique ID, and given instructions on how to collect the sample. They will return the sample to study staff, who will assess hydration on site and then dispose of the sample. If there is no latrine available on site, a private location where pupils provide a sample will be set up. Pupils will always be allowed to provide the sample alone. Study staff will provide water and soap for handwashing so pupils can wash their hands after giving the urine sample. In the morning, the urine sample will be collected immediately following the pupil interview. In the afternoon, the urine sample will be collected immediately prior to commencing cognitive testing.

Cognitive tests + self-report scales. Cognitive tests will be paper-based and will be administered in a group setting in the classroom by trained study enumerators. Schoolteachers and administrators will be asked to leave the classroom during the testing period. Each pupil will be provided with a booklet containing a set of cognitive tests and self- assessment scales of thirst, mood, and perceived difficulty. Cognitive tests and self- assessment scales will be administered once in the morning and once in the afternoon by study staff. Total testing time for the session is estimated to be a maximum of 45 minutes.

Hydration status measures

Hydration status will be measured through urinalysis using three methods: urine specific gravity, urine color, and self-reported thirst. The urine sample will be used assess urine specific gravity and color on site. Study staff will record measurements and then discard the sample. Pupils will self-report thirst twice on the day of testing (morning and afternoon) using a scale contained within the cognitive testing booklet.

Cognitive test performance measures

Cognitive performance will be assessed through a series of seven simple tests assessing a broad range of cognitive skills, adapted from past research that has been carried out in children in Israel and the United Kingdom. All cognitive assessments will be adapted specifically for the Mali context prior to data collection, and local enumerators will be trained on the administration of these tests. The investigators will collaborate with implementing partners to translate test instructions into local languages as needed and pre-test to ensure tools are appropriate for the study context. All tests will be paper-based tests and will be scored manually.

Risks to participation

There are minimal risks to participation in this study. The biggest risk of participation is lost class time. Participation in the study will not subject participants to any excess risk other than two interruptions of class time between 30-45 minutes each, a single interruption of 5 minutes to complete the individual interview, and the time it takes to provide a urine sample. All activities have been designed to minimize time taken away from class instruction, and all efforts will be made not to cause other disruptions. Study staff will ensure that head teachers, other teachers, and pupil participants all fully understand that performance on cognitive tests does not affect their grade, and that urine samples will be discarded.

Response booklets will be stored in a locked office, and data will be entered into a secure database. No personal identifying information will be kept with the data.

Benefits to subject or future benefits

The only direct benefit of participation in this study is that all participants will be provided with drinking water during one school day. There are no other direct benefits to participants other than knowing that information gained from this study will contribute to knowledge about the educational and health impacts of improved WASH in schools. The information will be shared with local stakeholders for potential use as an advocacy tool so that future programs in this and other areas can build upon the work that is done in this program.

Data analysis

Results from surveys, cognitive tests, and urine samples will be entered into a password-protected excel database. The database will be exported as the appropriate statistical analysis software file. Paired t-tests will be conducted to compare change in test score from baseline and follow-up between different groups (e.g., water vs. no water; dehydrated vs. hydrated).

Data management and monitoring

This trial does not entail a medical intervention of any kind; therefore, a typical data safety and monitoring plan is not necessary. Study staff will be instructed to monitor any unforeseen situations that suggest an increase in risk to participants and immediately inform the study manager so that a decision can be made on how to mitigate those risks.

Confidentiality

Pupils will be assigned a unique identifier at the start of data collection. Stickers with this identifier will be placed on all pupil testing materials. A list linking identifiers to pupils will be created to assist data collection logistics during the course of the data collection period; however, this list will be disposed of after the data collection period is ended. No personal identifying information will be collected as part of this study.

No personal identifiers will be kept in the database. All samples will be destroyed before leaving the study site and no samples will be banked as part of this study.

Informed Consent

A waiver of parental consent for pupil data collection will be secured from the government authority body such as the Ministry of Education.

In the local setting, a signed consent will also be obtained from the school management committee (SMC), or in its absence, from the school director. In Mali, the SMC is empowered to oversee management and activities at the school, on behalf of the community that school serves. At each school, the SMC chairperson or school director (as appropriate) will be asked to sign in loco parentis ("in the place of parent") on behalf of the pupil participants. The consent procedure will inform the school of the activities, purpose of the research, and will obtain permission for the researchers to carry out activities with assenting pupils.

School directors and SMC chairpersons would sign the in loco parentis form for up to 150 pupils at each school. This form will be signed at the first visit, and will serve as consent for all subsequent visits. One in loco parentis forms will be collected from each school, with up to four total being collected for this study (one for each of the four schools).

All pupil subjects in the classes selected to participate in the study will be read a complete informed oral assent script as a group prior to any data collection by a trained staff member. The staff member will then call the pupils outside of the class one by one and ask if they have any questions about the explanation that was given in class, and answer any questions they may have. They will then ask if the pupil assents, and record assent on the list of pupils. While the study will be explained to the class as a group, the actual pupil assent will be taken in this private setting so that there is no appearance of coercion from classmates or teachers.

Once a pupil assents, the study staff member will commence with the screening test. If the pupil passes the test, the study staff will administer the pupil questionnaire. Once the questionnaire is complete, the pupil will be given a collection cup and asked to provide a sample.

Oral assent has been chosen rather than written due to varying levels of literacy at the school as well as a desire to minimize paperwork that contains participants' names.

A maximum of 150 assents will be recorded at each study school, with a maximum of 300 total pupil assents recorded over the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Attend a school pre-selected for the study
* Attend grade level 3-6
* Understand and respond to verbal instruction

Exclusion Criteria:

* Unable to write down a string of numbers

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2013-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Cognitive test performance | 5-8 hours following intervention
  Measured by paper-based tests of visual attention, visual memory, short-term member, and visuomotor skills

SECONDARY OUTCOMES:
Perceived difficulty of task | 5-8 hours followign intervention
  Measured by self-report
Hydration status | 5-8 hours following intervention
  Measured by urine specific gravity,urine color, and self-reported thirst

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Freeman, PhD MPH, Principal Investigator — Emory University
Locations (1):
- Sikasso rural, Sikasso, Mali

REFERENCES:
- [Result] Chard AN, Trinies V, Edmonds CJ, Sogore A, Freeman MC. The impact of water consumption on hydration and cognition among schoolchildren: Methods and results from a crossover trial in rural Mali. PLoS One. 2019 Jan 17;14(1):e0210568. doi: 10.1371/journal.pone.0210568. eCollection 2019. PMID 30653554